CLINICAL TRIAL: NCT04384913
Title: Kinematic Versus Mechanical Alignment in Total Knee Replacement: a Randomized Double-blinded Controlled Study
Brief Title: Kinematic Versus Mechanical Alignment in Total Knee Replacement
Acronym: KAvsMA
Status: Active, not recruiting | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: A2-2017-KAvsMA
Record Dates: First submitted 2020-04-28; First posted 2020-05-12 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Total Knee Replacement
Keywords: TKA (Total knee arthroplasty); KA (kinematic alignment)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MA (mechanical alignment): Patients in group MA (mechanical alignment) will be operated according to mechanical implantation technique. In the mechanical group, femoral and tibial cutting blocks will be designed for a 0-degree angle according to the mechanical axis. Femoral rotation will be aligned with the femoral trans-epicondylar axis. Tibial rotation will follow femoral rotation.
- KA (kinematic alignment): Patients in group KA (kinematic alignment) will be operated according to kinematic implantation technique. The kinematic cutting blocks will be designed to resurface the femoral and tibial bones to restore each patient´s pre-arthritic anatomy and Joint line. Based on a available CT dat the prearthritic anatomy is reconstructed by compensating bone defects and restoring the physiological cartilage height of 1,7mm. Femoral Flexion is evaluated by the anterior Cortex of the distal femur, tibia slope is defined to 3° due to ACL (Anterior Cruciate Ligament) loss, but cab be adapted during surgery.

SUMMARY:
This prospective controlled double-blind randomized study compares kinematic and mechanical alignment in TKA (Total knee arthroplasty). A total of 120 patients will be included and the surgery will be performed using CT based 3D printed PSI(Patient Specific Instruments) Cutting guides.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is known, to significantly improve function and satisfaction in arthritic knee patients; nevertheless, a substantial percentage of these patients are not fully satisfied. Thus, several authors reported significantly improved outcomes after slightly under correcting varus knees after TKA. The concept of kinematic alignment (KA) even more addresses the patient´s individual anatomy with three-dimensional restoration of individual axes, joint lines and joint envelope of laxity. The aim of this prospective randomized study was to demonstrate equivalence between mechanical and kinematic alignment in restoring knee function in terms of subjective and objective outcomes.

In this prospective randomized controlled double-blind study 120 patients with osteoarthritic knees will be treated with a Medial Pivot TKA (Medacta Sphere GMK). The patients are divided into two groups. Group A receive the TKA using mechanical alignment principles, group B receive the kinematic alignment. The surgical technique was equal in both groups. CT-based 3D printed PSI cutting blocks were used for the saw cuts. Pre and postoperative standard x-rays were performed. To determine the subjective and objective outcomes the OKS(Oxford Knee Score), the KSS(Knee Society Sore), the FJS-12(Forgotten Joint Score) and the WOMAC Score were collected.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the knee
* Primary TKA
* UCLA Score (University of California, Los Angeles Score)>/= 4
* mMPTA: 85°- 90°
* Sum of mMPTA(mechanical medial proximal tibial angle) and mLDFA(mechanical lateral distal femoral angle) between 3°varus and 2°valgus from neutral

Exclusion Criteria:

* Minor Patient
* Pregnant or breast feeding woman
* Difference in the radius of medial and lateral condyles >2mm
* Previous osteotomy around the knee
* BMI >40
* Ligament instability likely to require higher level of constraint
* Previous infection or inflammatory disease
* Any Patient who cannot or will not provide informed consent for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Symptomatic osteoarthritis of the knee
  * Primary TKA
  * UCLA>/= 4
  * mMPTA: 85°- 90°
  * Sum of mMPTA and mLDFA between 3°varus and 2°valgus from neutral
  Exclusion Criteria:
  * Minor Patient
  * Pregnant or breast feeding woman
  * Difference in the radius of medial and lateral condyles >2mm
  * Previous osteotomy around the knee
  * BMI >40
  * Ligament instability likely to require higher level of constraint
  * Previous infection or inflammatory disease
  * Any Patient who cannot or will not provide informed consent for participation in the study
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score (KSS) | 3 months postoperative
  The Knee Society Scoring System is a validated and responsive method for assessing objective and subjective outcomes after total and partial knee arthroplasty.
  Minimum: 0 (worst), Maximum: 100 (best)
Knee Society Score (KSS) | 12 months postoperative
  The Knee Society Scoring System is a validated and responsive method for assessing objective and subjective outcomes after total and partial knee arthroplasty.
  Minimum: 0 (worst), Maximum: 100 (best)
Knee Society Score (KSS) | 24 months postoperative
  The Knee Society Scoring System is a validated and responsive method for assessing objective and subjective outcomes after total and partial knee arthroplasty.
  Minimum: 0 (worst), Maximum: 100 (best)

SECONDARY OUTCOMES:
Forgotten Joint Score (FJS-12) | 3 months postoperative
  The FJS Knee was designed to assess patient outcome in patients undergoing conservative or operative treatment of the knee. This questionnaire shows its strengths in patients with a good level of knee function and a low pain level. It has been designed specifically to reduce ceiling effects commonly associated with many PRO measures in this patient group, e.g. when assessing short- to mid-term results in total knee arthroplasty patients.
  Minimum: 0 (worst), Maximum: 100 (best)
Forgotten Joint Score (FJS-12) | 12 months postoperative
  The FJS Knee was designed to assess patient outcome in patients undergoing conservative or operative treatment of the knee. This questionnaire shows its strengths in patients with a good level of knee function and a low pain level. It has been designed specifically to reduce ceiling effects commonly associated with many PRO measures in this patient group, e.g. when assessing short- to mid-term results in total knee arthroplasty patients.
  Minimum: 0 (worst), Maximum: 100 (best)
Forgotten Joint Score (FJS-12) | 24 months postoperative
  The FJS Knee was designed to assess patient outcome in patients undergoing conservative or operative treatment of the knee. This questionnaire shows its strengths in patients with a good level of knee function and a low pain level. It has been designed specifically to reduce ceiling effects commonly associated with many PRO measures in this patient group, e.g. when assessing short- to mid-term results in total knee arthroplasty patients.
  Minimum: 0 (worst), Maximum: 100 (best)
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 3 months postoperative
  The WOMAC Score was developed in 1982 and is a Patient Reported Outcome (PRO) instrument to assess the effects of osteoarthritis of the hip and/or knee joint in affected patients. The WOMAC-Score contains 24 questions and is able to assess the effects of osteoarthritis of the hip and/or knee joint with regard to three subscales:
  Pain - 5 questions Stiffness - 2 questions Physical function - 17 questions Minimum: 0 (best), Maximum: 100 (worst)
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 12 months postoperative
  The WOMAC Score was developed in 1982 and is a Patient Reported Outcome (PRO) instrument to assess the effects of osteoarthritis of the hip and/or knee joint in affected patients. The WOMAC-Score contains 24 questions and is able to assess the effects of osteoarthritis of the hip and/or knee joint with regard to three subscales:
  Pain - 5 questions Stiffness - 2 questions Physical function - 17 questions Minimum: 0 (best), Maximum: 100 (worst)
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 24 months postoperative
  The WOMAC Score was developed in 1982 and is a Patient Reported Outcome (PRO) instrument to assess the effects of osteoarthritis of the hip and/or knee joint in affected patients. The WOMAC-Score contains 24 questions and is able to assess the effects of osteoarthritis of the hip and/or knee joint with regard to three subscales:
  Pain - 5 questions Stiffness - 2 questions Physical function - 17 questions Minimum: 0 (best), Maximum: 100 (worst)
Oxford Knee Score (OKS) | 3 months postoperative
  The OKS questionnaire consists of 12 questions that cover function and pain of the knee. Each question is scored from 0 to 4 (0 being the worst outcome and 4 being the best). The overall score is the sum of all items and can range from 0 to 48, with higher scores corresponding to better outcomes. The OKS has a big ceiling effect and cannot differentiate between good and very good results. However, the most of the researchers world wide use the OKS as a reference.
Oxford Knee Score (OKS) | 12 months postoperative
  The OKS questionnaire consists of 12 questions that cover function and pain of the knee. Each question is scored from 0 to 4 (0 being the worst outcome and 4 being the best). The overall score is the sum of all items and can range from 0 to 48, with higher scores corresponding to better outcomes. The OKS has a big ceiling effect and cannot differentiate between good and very good results. However, the most of the researchers world wide use the OKS as a reference.
Oxford Knee Score (OKS) | 24 months postoperative
  The OKS questionnaire consists of 12 questions that cover function and pain of the knee. Each question is scored from 0 to 4 (0 being the worst outcome and 4 being the best). The overall score is the sum of all items and can range from 0 to 48, with higher scores corresponding to better outcomes. The OKS has a big ceiling effect and cannot differentiate between good and very good results. However, the most of the researchers world wide use the OKS as a reference.

CONTACTS AND LOCATIONS:
Overall Officials: Max Ettinger, Prof. Dr., Principal Investigator — Orthopädische Klinik der Medizinischen Hochschule Hannover im DIAKOVERE Annastift
Locations (1):
- Orthopädische Klinik der Medizinischen Hochschule Hannover im DIAKOVERE Annastift, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No